CLINICAL TRIAL: NCT01308580
Title: Randomized, Open Label Multi-Center Study Comparing Cabazitaxel at 20 mg/m² and at 25 mg/m² Every 3 Weeks in Combination With Prednisone for the Treatment of Metastatic Castration Resistant Prostate Cancer Previously Treated With a Docetaxel-Containing Regimen
Brief Title: Cabazitaxel at 20 mg/m² Compared to 25 mg/m² With Prednisone for the Treatment of Metastatic Castration Resistant Prostate Cancer
Acronym: PROSELICA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC11785; 2010-022163-35 (EudraCT Number)
Record Dates: First submitted 2011-03-03; First posted 2011-03-04 (Estimated); Results first posted 2016-10-11 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2016-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cabazitaxel; XRP6258; Prednisone; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cabazitaxel 20 mg/m^2 (Experimental): Cabazitaxel 20 mg/m^2 intravenous (IV) infusion over 1 hour on Day 1 of each 21-day cycle in combination with Prednisone (or Prednisolone) 10 mg orally daily until disease progression (DP), unacceptable toxicity, participant's refusal of further study treatment or for a maximum of 10 cycles.
  Interventions: Drug: Cabazitaxel (XRP6258); Drug: Prednisone (or Prednisolone)
- Cabazitaxel 25 mg/m^2 (Experimental): Cabazitaxel 25 mg/m^2 IV infusion over 1 hour on Day 1 of each 21-day cycle in combination with Prednisone (or Prednisolone) 10 mg orally daily until DP, unacceptable toxicity, participant's refusal of further study treatment or for a maximum of 10 cycles.
  Interventions: Drug: Cabazitaxel (XRP6258); Drug: Prednisone (or Prednisolone)

INTERVENTIONS:
Drug: Cabazitaxel (XRP6258) — Pharmaceutical form: Concentrate and solvent for solution for infusion
  Route of administration: Intravenous
  Other Names: Jevtana®
Drug: Prednisone (or Prednisolone) — Pharmaceutical form: Tablet
  Route of administration: Oral

SUMMARY:
Primary Objective:

- To demonstrate the non inferiority in term of overall survival (OS) of Cabazitaxel 20 mg/m² (Arm A) versus Cabazitaxel 25 mg/m² (Arm B) in combination with prednisone in participants with metastatic castration resistant prostate cancer (mCRPC) previously treated with a docetaxel-containing regimen.

Secondary Objectives:

* To evaluate safety in the 2 treatment arms and to assess if Cabazitaxel 20 mg/m² was better tolerated than Cabazitaxel 25 mg/m².
* To compare efficacy of Cabazitaxel at 20 mg/m² and 25 mg/m² for:

  * Progression Free Survival (PFS) defined as the first occurrence of any of the following events: tumor progression per Response Evaluation Criteria In Solid Tumors (RECIST), prostate-specific antigen (PSA) progression, pain progression or death due to any cause;
  * PSA Progression;
  * Pain progression;
  * Tumor response in participants with measurable disease (RECIST 1.1);
  * PSA response;
  * Pain response in participants with stable pain at baseline.
* To compare Health-related Quality of Life (HRQoL).
* To assess the pharmacokinetics and pharmacogenomics of Cabazitaxel.

DETAILED DESCRIPTION:
Participants were treated until DP, unacceptable toxicity, participant's refusal of further study treatment or for a maximum of 10 cycles. All participants were followed when on study treatment and after completion of study treatment during follow up period until death or the study cutoff date, whichever came first.

ELIGIBILITY:
Inclusion criteria :

I 01. Diagnosis of histologically or cytologically proven prostate adenocarcinoma, that was resistant to hormone therapy and previously treated with a docetaxel-containing regimen.

I 02. Participant must had either measurable or non-measurable disease. I 03. Received prior castration by orchiectomy and/or Luteinizing Hormone-Releasing Hormone (LH-RH) agonist with or without antiandrogen, antiandrogen withdrawal, monotherapy with estramustine, or other hormonal agents.

I 04. Life expectancy > 6 months. I 05. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 - 2 (i.e, participant must be ambulatory, capable of all self-care, and up and about more than 50% of waking hours).

I 06. Age ≥18 years (or country's legal age of majority if the legal age was > 18 years).

Exclusion criteria:

E 01. Previous treatment with mitoxantrone or cabazitaxel. E 02. Prior isotope therapy or radiotherapy to ≥30% of bone marrow. In case of prior isotope therapy 12 weeks must had elapsed prior to first study drug administration.

E 03. Adverse events (excluding alopecia and those listed in the specific exclusion criteria) from any prior anticancer therapy of grade >1(National Cancer Institute Common Terminology Criteria [NCI CTCAE] v4.03) at the time of randomization.

E 04. Prior surgery, radiation, chemotherapy, or other anti-cancer therapy within 4 weeks prior to enrollment in the study.

E 05. Prior malignancy. Adequately treated basal cell or squamous cell skin or superficial (pTis, pTa, and pT1) bladder cancer were allowed, as well as any other cancer for which chemotherapy had been completed ≥ 5 years ago and from which the participant had been disease-free for ≥ 5 years.

E 06. Participation in another clinical trial and any concurrent treatment with any investigational drug within 30 days prior to randomization.

E 07. Known brain or leptomeningeal involvement. E 08. Other concurrent serious illness or medical conditions. E 09. Uncontrolled cardiac arrhythmias, angina pectoris, and/or hypertension. History of congestive heart failure (NYHA III or IV) or myocardial infarction within last 6 months was also not allowed.

E 10. Any severe acute or chronic medical condition which could impair the ability of the participant to participate to the study or to comply with the study procedures or interfere with interpretation of study results.

E 11. Absence of signed and dated Institutional Review Board (IRB)-approved participant informed consent form prior to enrollment into the study.

E 12. Participants with reproductive potential who did not agree to use accepted and effective method of contraception during the study treatment period. The definition of "effective method of contraception" was based on the Investigator's judgment. Participant's Partners of childbearing potential (unless surgically sterile, post menopausal or for another reason had no chance of becoming pregnant) not protected by highly effective contraceptive method of birth control as defined for contraception in the Informed Consent Form and /or in a local protocol addendum.

E 13. History of hypersensitivity to docetaxel, or polysorbate 80. E 14. Inadequate organ and bone marrow function. E 15. Contraindications to the use of corticosteroid treatment. E 16. Symptomatic peripheral neuropathy grade > 2 (NCI CTCAE v.4.03).

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2011-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (172):
- United States (21):
  - Investigational Site Number 840002, Muscle Shoals, Alabama
  - Investigational Site Number 840004, Hot Springs, Arkansas
  - Investigational Site Number 840008, Anaheim, California
  - Investigational Site Number 840010, La Jolla, California
  - Investigational Site Number 840001, San Bernardino, California
  - Investigational Site Number 840021, Stamford, Connecticut
  - Investigational Site Number 840023, Jacksonville, Florida
  - Investigational Site Number 840013, Lakeland, Florida
  - Investigational Site Number 840003, Port Saint Lucie, Florida
  - Investigational Site Number 840007, New Orleans, Louisiana
  - Investigational Site Number 840014, Baltimore, Maryland
  - Investigational Site Number 840005, Rockville, Maryland
  - Investigational Site Number 840017, Saint Louis Park, Minnesota
  - Investigational Site Number 840011, Jackson, Mississippi
  - Investigational Site Number 840016, Lincoln, Nebraska
  - Investigational Site Number 840015, East Orange, New Jersey
  - Investigational Site Number 840024, Raleigh, North Carolina
  - Investigational Site Number 840020, Akron, Ohio
  - Investigational Site Number 840006, Pawtucket, Rhode Island
  - Investigational Site Number 840025, Chattanooga, Tennessee
  - Investigational Site Number 840012, Corpus Christi, Texas
- Argentina (4):
  - Investigational Site Number 032002, Buenos Aires
  - Investigational Site Number 032001, Rosario
  - Investigational Site Number 032003, Salta
  - Investigational Site Number 032004, Santa Fe
- Australia (15):
  - Investigational Site Number 036014, Adelaide
  - Investigational Site Number 036013, Bankstown
  - Investigational Site Number 036010, Box Hill
  - Investigational Site Number 036012, Camperdown
  - Investigational Site Number 036008, Coffs Harbour
  - Investigational Site Number 036001, Concord
  - Investigational Site Number 036015, Elizabeth Vale
  - Investigational Site Number 036009, Fitzroy
  - Investigational Site Number 036007, Garran
  - Investigational Site Number 036005, Heidelberg West
  - Investigational Site Number 036002, Malvern
  - Investigational Site Number 036006, South Brisbane
  - Investigational Site Number 036016, Subiaco
  - Investigational Site Number 036003, Wahroonga
  - Investigational Site Number 036004, Wodonga
- Belgium (14):
  - Investigational Site Number 056007, Antwerp
  - Investigational Site Number 056001, Brussels
  - Investigational Site Number 056008, Brussels
  - Investigational Site Number 056002, Brussels
  - Investigational Site Number 056009, Charleroi
  - Investigational Site Number 056003, Ghent
  - Investigational Site Number 056012, Godinne
  - Investigational Site Number 056016, Haine-Saint-Paul
  - Investigational Site Number 056005, Hasselt
  - Investigational Site Number 056010, Libramont
  - Investigational Site Number 056013, Liège
  - Investigational Site Number 056011, Ottignies
  - Investigational Site Number 056004, Roeselare
  - Investigational Site Number 056006, Turnhout
- Brazil (12):
  - Investigational Site Number 076016, Fortaleza
  - Investigational Site Number 076012, Ijuí
  - Investigational Site Number 076015, Mogi das Cruzes
  - Investigational Site Number 076014, Porto Alegre
  - Investigational Site Number 076010, Rio de Janeiro
  - Investigational Site Number 076007, Salvador
  - Investigational Site Number 076003, São José do Rio Preto
  - Investigational Site Number 076009, São Paulo
  - Investigational Site Number 076001, São Paulo
  - Investigational Site Number 076013, São Paulo
  - Investigational Site Number 076008, São Paulo
  - Investigational Site Number 076002, São Paulo
- Canada (4):
  - Investigational Site Number 124002, Greenfield Park
  - Investigational Site Number 124001, Oshawa
  - Investigational Site Number 124003, Ottawa
  - Investigational Site Number 124005, Owen Sound
- Chile (4):
  - Investigational Site Number 152005, Santiago
  - Investigational Site Number 152004, Santiago
  - Investigational Site Number 152002, Santiago
  - Investigational Site Number 152001, Viña del Mar
- France (11):
  - Investigational Site Number 250005, Avignon
  - Investigational Site Number 250008, Hyères
  - Investigational Site Number 250001, La Roche-sur-Yon
  - Investigational Site Number 250002, Nantes
  - Investigational Site Number 250004, Nîmes
  - Investigational Site Number 250010, Paris
  - Investigational Site Number 250009, Reims
  - Investigational Site Number 250007, Reims
  - Investigational Site Number 250006, Saint-Brieuc
  - Investigational Site Number 250003, Toulouse
  - Investigational Site Number 250011, Toulouse
- Germany (11):
  - Investigational Site Number 276003, Aachen
  - Investigational Site Number 276007, Dresden
  - Investigational Site Number 276004, Düsseldorf
  - Investigational Site Number 276001, Erlangen
  - Investigational Site Number 276011, Hamburg
  - Investigational Site Number 276005, Hamburg
  - Investigational Site Number 276010, Homburg
  - Investigational Site Number 276006, München
  - Investigational Site Number 276012, Nürtingen
  - Investigational Site Number 276008, Tübingen
  - Investigational Site Number 276002, Wuppertal
- Hungary (5):
  - Investigational Site Number 348001, Budapest
  - Investigational Site Number 348005, Budapest
  - Investigational Site Number 348004, Budapest
  - Investigational Site Number 348006, Miskolc
  - Investigational Site Number 348003, Pécs
- Netherlands (5):
  - Investigational Site Number 528005, Arnhem
  - Investigational Site Number 528003, Blaricum
  - Investigational Site Number 528004, Hoofddorp
  - Investigational Site Number 528002, Nijmegen
  - Investigational Site Number 528001, Zwolle
- Peru (7):
  - Investigational Site Number 604003, Arequipa
  - Investigational Site Number 604006, Lima
  - Investigational Site Number 604001, Lima
  - Investigational Site Number 604007, Lima
  - Investigational Site Number 604002, Lima
  - Investigational Site Number 604004, Lima
  - Investigational Site Number 604005, Lima
- Poland (5):
  - Investigational Site Number 616006, Lubin
  - Investigational Site Number 616002, Olsztyn
  - Investigational Site Number 616001, Rybnik
  - Investigational Site Number 616005, Siedlce
  - Investigational Site Number 616004, Torun
- Romania (11):
  - Investigational Site Number 642005, Alba Iulia
  - Investigational Site Number 642006, Baia Mare
  - Investigational Site Number 642009, Bucharest
  - Investigational Site Number 642008, Bucharest
  - Investigational Site Number 642001, Cluj-Napoca
  - Investigational Site Number 642003, Cluj-Napoca
  - Investigational Site Number 642004, Cluj-Napoca
  - Investigational Site Number 642002, Cluj-Napoca
  - Investigational Site Number 642012, Focşani
  - Investigational Site Number 642007, Hunedoara
  - Investigational Site Number 642013, Onești
- Russia (9):
  - Investigational Site Number 643007, Moscow
  - Investigational Site Number 643005, Moscow
  - Investigational Site Number 643004, Moscow
  - Investigational Site Number 643006, Moscow
  - Investigational Site Number 643008, Obninsk
  - Investigational Site Number 643001, Saint Petersburg
  - Investigational Site Number 643010, Saint Petersburg
  - Investigational Site Number 643003, Tula
  - Investigational Site Number 643009, Yekaterinburg
- South Africa (5):
  - Investigational Site Number 710003, Cape Town
  - Investigational Site Number 710002, Durban
  - Investigational Site Number 710005, Johannesburg
  - Investigational Site Number 710004, Johannesburg
  - Investigational Site Number 710001, Pretoria
- South Korea (5):
  - Investigational Site Number 410003, Seongnam
  - Investigational Site Number 410002, Seoul
  - Investigational Site Number 410004, Seoul
  - Investigational Site Number 410005, Seoul
  - Investigational Site Number 410001, Seoul
- Spain (8):
  - Investigational Site Number 724003, Badalona
  - Investigational Site Number 724001, Barcelona
  - Investigational Site Number 724002, Madrid
  - Investigational Site Number 724008, Madrid
  - Investigational Site Number 724006, Málaga
  - Investigational Site Number 724005, Palma de Mallorca
  - Investigational Site Number 724004, Sabadell
  - Investigational Site Number 724007, Seville
- Taiwan (3):
  - Investigational Site Number 158002, Taiching
  - Investigational Site Number 158003, Tainan
  - Investigational Site Number 158001, Taipei
- Tunisia (3):
  - Investigational Site Number 788004, Sfax
  - Investigational Site Number 788003, Sousse
  - Investigational Site Number 788002, Tunis
- Turkey (Türkiye) (3):
  - Investigational Site Number 792003, Antalya
  - Investigational Site Number 792001, Bornova
  - Investigational Site Number 792002, Istanbul
- United Kingdom (7):
  - Investigational Site Number 826002, Birmingham
  - Investigational Site Number 826004, Colchester
  - Investigational Site Number 826005, Glasgow
  - Investigational Site Number 826006, Guildford
  - Investigational Site Number 826007, Manchester
  - Investigational Site Number 826003, Newcastle upon Tyne
  - Investigational Site Number 826001, Sutton

REFERENCES:
- [Derived] Meisel A, de Wit R, Oudard S, Sartor O, Stenner-Liewen F, Shun Z, Foster M, Ozatilgan A, Eisenberger M, de Bono JS. Neutropenia, neutrophilia, and neutrophil-lymphocyte ratio as prognostic markers in patients with metastatic castration-resistant prostate cancer. Ther Adv Med Oncol. 2022 Jun 1;14:17588359221100022. doi: 10.1177/17588359221100022. eCollection 2022. PMID 35677318
- [Derived] Thiery-Vuillemin A, Fizazi K, Sartor O, Oudard S, Bury D, Thangavelu K, Ozatilgan A, Poole EM, Eisenberger M, de Bono J. An analysis of health-related quality of life in the phase III PROSELICA and FIRSTANA studies assessing cabazitaxel in patients with metastatic castration-resistant prostate cancer. ESMO Open. 2021 Apr;6(2):100089. doi: 10.1016/j.esmoop.2021.100089. Epub 2021 Mar 16. PMID 33740734
- [Derived] Mehra N, Dolling D, Sumanasuriya S, Christova R, Pope L, Carreira S, Seed G, Yuan W, Goodall J, Hall E, Flohr P, Boysen G, Bianchini D, Sartor O, Eisenberger MA, Fizazi K, Oudard S, Chadjaa M, Mace S, de Bono JS. Plasma Cell-free DNA Concentration and Outcomes from Taxane Therapy in Metastatic Castration-resistant Prostate Cancer from Two Phase III Trials (FIRSTANA and PROSELICA). Eur Urol. 2018 Sep;74(3):283-291. doi: 10.1016/j.eururo.2018.02.013. Epub 2018 Feb 28. PMID 29500065
- [Derived] Eisenberger M, Hardy-Bessard AC, Kim CS, Geczi L, Ford D, Mourey L, Carles J, Parente P, Font A, Kacso G, Chadjaa M, Zhang W, Bernard J, de Bono J. Phase III Study Comparing a Reduced Dose of Cabazitaxel (20 mg/m2) and the Currently Approved Dose (25 mg/m2) in Postdocetaxel Patients With Metastatic Castration-Resistant Prostate Cancer-PROSELICA. J Clin Oncol. 2017 Oct 1;35(28):3198-3206. doi: 10.1200/JCO.2016.72.1076. Epub 2017 Aug 15. PMID 28809610
- [Derived] Winquist E, Rodrigues G. Open clinical uro-oncology trials in Canada. Can J Urol. 2012 Dec;19(6):6587-91. No abstract available. PMID 23228299

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 172 centers in 22 countries. A total of 1463 participants were screened between 19 April 2011 and 18 November 2013. Out of 1463 participants, 1200 participants were enrolled in this study and 263 were not eligible to join the study.
Pre-assignment Details: Participants were randomized by Interactive Voice Response System (IVRS) in 1:1 ratio (Cabazitaxel 20 mg/m^2: Cabazitaxel 25 mg/m^2) and stratified according to Eastern Cooperative Oncology Group Performance Status (ECOG PS) score (0 or 1 versus 2), measurability of disease (measurable versus non-measurable) and region.
Period: Overall Study
Arm/Group | Cabazitaxel 20 mg/m^2 | Cabazitaxel 25 mg/m^2
Started | 598 | 602
Treated | 587 (Random assignment, was not actual treatment in some cases) | 588 (Random assignment, was not actual treatment in some cases)
Completed | 586 (Completed participants included those who withdrew treatment consent but were followed for survival) | 595 (Completed participants included those who withdrew treatment consent but were followed for survival)
Not Completed | 12 | 7
Not completed — Lost to Follow-up | 12 | 7

BASELINE CHARACTERISTICS:
Groups:
- Cabazitaxel 20 mg/m^2: Cabazitaxel 20 mg/m^2 IV infusion over 1 hour on Day 1 of each 21-day cycle in combination with Prednisone (or Prednisolone) 10 mg orally daily until DP, unacceptable toxicity, participant's refusal of further study treatment or for a maximum of 10 cycles.
- Total: Total of all reporting groups
Arm/Group | Cabazitaxel 20 mg/m^2 | Cabazitaxel 25 mg/m^2 | Total
Number analyzed (Participants) | 598 | 602 | 1200
Age, Customized [Number; unit: participants]
  <65 years | 182 | 180 | 362
  65 to 74 years | 296 | 295 | 591
  ≥75 years | 120 | 127 | 247
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 598 | 602 | 1200

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time interval from the date of randomization to the date of death due to any cause. In absence of confirmation of death, survival time was censored at the earlier of the last date the participant was known to be alive or the study cut-off date. The cut-off date for the final analysis of OS was the date when the 988th death had been observed. Analysis was performed by Kaplan-Meier method.
Time Frame: From baseline up to death due to any cause or study cut-off date, whichever was earlier (maximum duration: 48 months)
Population: Analysis was performed on Intent-to-Treat (ITT) population, which included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabazitaxel 20 mg/m^2 | Cabazitaxel 25 mg/m^2
Number analyzed (Participants) | 598 | 602
months | 13.4 [12.19 to 14.88] | 14.5 [13.47 to 15.28]
Statistical Analysis 1: Comparison: Cabazitaxel 20 mg/m^2 vs Cabazitaxel 25 mg/m^2; The hazard ratio for OS was estimated using the Cox proportional hazards regression model. The Cox proportional hazard model was adjusted by measurability of the disease at baseline, ECOG PS score at baseline, and region at the time of randomization. Cabazitaxel 20 mg/m^2 relative to 25 mg/m^2 dose group was considered non-inferior if the upper bound of 1-sided 98.89% confidence interval of hazard ratio (20 mg/m^2 versus 25 mg/m^2) was less than the non-inferiority margin of 1.214; Test type: Non-Inferiority or Equivalence — Non-inferiority margin of 1.214; Hazard Ratio (HR) = 1.024, 98.89% CI 1-sided [upper limit 1.184] — Cabazitaxel 20 mg/m^2 vs Cabazitaxel 25 mg/m^2
Statistical Analysis 2: Comparison: Cabazitaxel 20 mg/m^2 vs Cabazitaxel 25 mg/m^2; The hazard ratio for OS was estimated using the Cox proportional hazards regression model. The Cox proportional hazard model was adjusted by measurability of the disease at baseline, ECOG PS score at baseline, and region at the time of randomization. Cabazitaxel 25 mg/m^2 was considered to be superior to 20 mg/m^2 dose if the lower bound of 1-sided 95% confidence interval of hazard ratio was greater than 1; Test type: Superiority or Other; Hazard Ratio (HR) = 1.024, 95% CI 1-sided [lower limit 0.922] — Cabazitaxel 20 mg/m^2 vs Cabazitaxel 25 mg/m^2

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was evaluated from date of randomization to date of first documentation of any of the events: 1) Radiological tumor progression: as per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1: at least a 20% increase in sum of diameters of target lesions (sum must also demonstrate an absolute increase of ≥5 mm) taking as reference the smallest sum while on study, appearance of one or more new lesions, or unequivocal progression of existing non target lesions, 2) Prostate Specific Antigen (PSA) progression: ≥25% increase over baseline/nadir value if baseline PSA ≥10 ng/mL; or 25% increase above the baseline level if baseline PSA >0 ng/mL & <10 ng/mL; or post-baseline value of >=2 ng/mL, if baseline PSA=0 ng/mL, 3) Pain progression: increase of ≥1 point in median Present Pain Intensity (PPI) from nadir or ≥25% increase in mean analgesic score (AS) from baseline score or requirement of local palliative radiotherapy, 4) Death. Analysis was performed by Kaplan-Meier method.
Time Frame: From baseline up to tumor progression, PSA progression, pain progression, death due to any cause or study cut-off date, whichever was earlier (maximum duration: 48 months)
Population: Analysis was performed on ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabazitaxel 20 mg/m^2 | Cabazitaxel 25 mg/m^2
Number analyzed (Participants) | 598 | 602
months | 2.9 [2.79 to 3.45] | 3.5 [3.12 to 3.94]
Statistical Analysis 1: Comparison: Cabazitaxel 20 mg/m^2 vs Cabazitaxel 25 mg/m^2; Hazard ratio was estimated using a Cox Proportional Hazards regression model. The Cox proportional hazard model was adjusted by measurability of the disease at baseline, ECOG PS score at baseline, and region at the time of randomization; Test type: Superiority or Other; Hazard Ratio (HR) = 1.099, 95% CI 2-sided [0.974 to 1.24] — Cabazitaxel 20 mg/m^2 vs Cabazitaxel 25 mg/m^2

3. Secondary Outcome: Time to Tumor Progression
Description: Time to Tumor progression was defined as the first occurrence of radiological tumor progression according to RECIST 1.1. Radiological tumor progression was defined at least a 20% increase in sum of diameters of target lesions (sum must also demonstrate an absolute increase of ≥5 mm) taking as reference the smallest sum while on study, appearance of one or more new lesions, or unequivocal progression of existing non target-lesions. Analysis was performed by Kaplan-Meier method.
Time Frame: From baseline up to tumor progression or death due to any cause or study cut-off date, whichever was earlier (maximum duration: 48 months)
Population: Analysis was performed on ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabazitaxel 20 mg/m^2 | Cabazitaxel 25 mg/m^2
Number analyzed (Participants) | 598 | 602
months | 9.0 [8.38 to 9.79] | 9.3 [8.61 to 9.92]
Statistical Analysis 1: Comparison: Cabazitaxel 20 mg/m^2 vs Cabazitaxel 25 mg/m^2; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Hazard Ratio (HR) = 1.096, 95% CI 2-sided [0.902 to 1.331] — Cabazitaxel 20 mg/m^2 vs Cabazitaxel 25 mg/m^2

4. Secondary Outcome: Percentage of Participants With Overall Objective Tumor Response
Description: Overall objective tumor response was defined as either a partial response (PR) or complete response (CR) according to the RECIST 1.1 criteria, as assessed by the investigator. CR was defined as disappearance of all target and non-target lesions and normalization of tumor marker level. Any pathological lymph nodes (whether target or non-target) must had reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From baseline up to DP or death due to any cause or study cut-off date, whichever was earlier (maximum duration: 48 months)
Population: Analysis was performed on ITT population. Number of participants analyzed= participants evaluable for tumor response with measurable disease at baseline and at least one valid post-baseline value.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cabazitaxel 20 mg/m^2 | Cabazitaxel 25 mg/m^2
Number analyzed (Participants) | 271 | 256
percentage of participants | 18.5 [13.8 to 23.1] | 23.4 [18.2 to 28.6]

5. Secondary Outcome: Time to PSA Progression
Description: Time to PSA progression was time interval between randomization & first occurrence of PSA progression. PSA progression defined as: 1) PSA responders (>50% decline from baseline PSA ≥10 ng/mL): increase of ≥25% (≥2 ng/mL) over nadir value, confirmed by second PSA ≥3 weeks later; 2) PSA non-responders (did not achieve >50% decline from baseline PSA ≥10 ng/mL): increase of ≥25% (≥2 ng/mL) over baseline value, confirmed by second PSA ≥3 weeks later; 3) In participants not eligible for PSA response (baseline PSA <10 ng/mL): (a) participants with baseline PSA >0 ng/mL & <10 ng/mL: increase in PSA by 25% (≥2 ng/mL) above baseline level, confirmed by second PSA value ≥3 weeks apart; (b) participants with baseline value=0 ng/mL: post-baseline PSA value ≥2 ng/mL. Note (for 1-3): Rise in PSA in first 12 weeks was progression only if met definition above and was associated with other sign of DP or if it continued beyond 12 weeks. Analysis was performed by Kaplan-Meier method.
Time Frame: From baseline up to PSA progression or death due to any cause or study cut-off date, whichever was earlier (maximum duration: 48 months)
Population: Analysis was performed on ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabazitaxel 20 mg/m^2 | Cabazitaxel 25 mg/m^2
Number analyzed (Participants) | 598 | 602
months | 5.7 [4.96 to 6.47] | 6.8 [6.11 to 7.46]
Statistical Analysis 1: Comparison: Cabazitaxel 20 mg/m^2 vs Cabazitaxel 25 mg/m^2; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Hazard Ratio (HR) = 1.195, 95% CI 2-sided [1.025 to 1.393] — Cabazitaxel 20 mg/m^2 vs Cabazitaxel 25 mg/m^2

6. Secondary Outcome: Percentage of Participants With PSA Response
Description: PSA response was defined as ≥50% decrease from baseline in serum PSA levels, confirmed by a second PSA value at least 3 weeks later in participants with baseline PSA value ≥10 ng/mL.
Time Frame: as for outcome 5
Population: Analysis was performed on ITT population. Number of participants analyzed= participants evaluable for PSA response with PSA value ≥10 ng/mL at baseline and at least one valid post-baseline value.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cabazitaxel 20 mg/m^2 | Cabazitaxel 25 mg/m^2
Number analyzed (Participants) | 543 | 538
percentage of participants | 29.5 [25.6 to 33.3] | 42.9 [38.8 to 47.1]

7. Secondary Outcome: Time to Pain Progression
Description: Pain Progression was defined as an increase of ≥1 point in the median PPI from its nadir confirmed by a second assessment at least 3 weeks later or ≥25 % increase in the mean AS compared with the baseline score confirmed by a second assessment at least 3 weeks later or requirement for local palliative radiotherapy. PPI was rated by participant in a diary using a scale of 0=no pain, 1=mild, 2=discomforting, 3=distressing, 4=horrible 5=excruciating. Analgesic use was recorded by the participant in a diary. AS was calculated from the analgesic use data based on a table of analgesic medications, with non-narcotic medications assigned a value of 1 point and narcotic medications assigned a value of 4 points. Analysis was performed by Kaplan-Meier method.
Time Frame: From baseline until DP, start of another anti-cancer therapy, death or study cut-off date (maximum duration: 48 months)
Population: Analysis was performed on ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabazitaxel 20 mg/m^2 | Cabazitaxel 25 mg/m^2
Number analyzed (Participants) | 598 | 602
months | 6.2 [5.22 to 7.39] | 6.4 [5.55 to 7.26]
Statistical Analysis 1: Comparison: Cabazitaxel 20 mg/m^2 vs Cabazitaxel 25 mg/m^2; Hazard ratio is estimated using a Cox Proportional Hazards regression model. The Cox proportional hazard model was adjusted by measurability of the disease at baseline, ECOG PS score at baseline, and region at the time of randomization; Test type: Superiority or Other; Hazard Ratio (HR) = 1.046, 95% CI 2-sided [0.874 to 1.251] — Cabazitaxel 20 mg/m^2 vs Cabazitaxel 25 mg/m^2

8. Secondary Outcome: Percentage of Participants With Pain Response
Description: Pain response was defined as either a ≥2-point decrease from baseline median PPI score without increase in AS, or a ≥50% decrease from baseline mean AS without increase in the PPI score, maintained for 2 consecutive evaluations at least 3 weeks apart. Increases in pain during the first 12 weeks were ignored in determining pain response.
Time Frame: From baseline until DP, start of another anti-cancer therapy, death or study cut-off date (maximum duration: 48 months)
Population: Analysis was performed on ITT population. Number of participants analyzed= participants evaluable for pain response with pain score with median PPI ≥2 and/or mean AS ≥10 points at baseline and at least one valid post-baseline value.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cabazitaxel 20 mg/m^2 | Cabazitaxel 25 mg/m^2
Number analyzed (Participants) | 248 | 284
percentage of participants | 34.7 [28.8 to 40.6] | 37.3 [31.7 to 42.9]

9. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-Prostate (FACT-P):Trial Outcome Index (TOI) as a Measure of Health Related Quality of Life (HRQoL)
Description: FACT-P is a 39-item participant questionnaire that measures the concerns of participants with prostate cancer. It consists of 5 sub-scales assessing physical well-being (7 items), social/family well-being (7 items), emotional well-being (6 items), functional well-being (7 items), and prostate-specific concerns (12 items). FACT-P TOI combines physical well-being, functional well-being, and prostate-specific concerns sub-scales for a total possible score range of 0 to 104, where higher values represent better HRQoL.
Time Frame: Baseline, Day 1 of each Cycle 1, 2, 3, 4, 5, 6, 7, 8, 9 and 10 (each cycle 21-day); post-treatment follow up 1 (up to 12 weeks)
Population: FACT-P population included randomized participants who completed FACT-P questionnaire at baseline & in at least one post-baseline assessment. Number of participants analyzed=participants with evaluable FACT-P TOI for specified outcome measure. Here, 'n' signifies number of participants with available data for specified category.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Cabazitaxel 20 mg/m^2 | Cabazitaxel 25 mg/m^2
Number analyzed (Participants) | 521 | 494
units on a scale
  Change from baseline at cycle 1 (n =521, 494) | 4.69 [2.95 to 6.44] | 5.08 [3.32 to 6.84]
  Change from baseline at cycle 2 (n = 500, 494) | 4.4 [2.67 to 6.14] | 5.55 [3.81 to 7.3]
  Change from baseline at cycle 3 (n =456, 451) | 3.75 [2 to 5.5] | 5.46 [3.7 to 7.23]
  Change from baseline at cycle 4 (n =420, 415) | 2.57 [0.8 to 4.33] | 3.82 [2.04 to 5.6]
  Change from baseline at cycle 5 (n =339, 361) | 1.78 [-0.03 to 3.59] | 3.06 [1.26 to 4.87]
  Change from baseline at cycle 6 (n =275, 318) | 2.57 [0.72 to 4.43] | 2.03 [0.2 to 3.86]
  Change from baseline at cycle 7 (n =225, 262) | 2.51 [0.6 to 4.42] | 2.73 [0.85 to 4.6]
  Change from baseline at cycle 8 (n =196, 227) | 1.44 [-0.5 to 3.39] | 2.08 [0.16 to 3.99]
  Change from baseline at cycle 9 (n =165, 172) | 0.94 [-1.06 to 2.94] | 1.46 [-0.55 to 3.46]
  Change from baseline at cycle 10 (n =137, 141) | 0.02 [-2.05 to 2.1] | 1.31 [-0.76 to 3.39]
  Change from baseline at Follow-up 1 (n =136, 152) | -2.27 [-4.35 to -0.19] | -1.16 [-3.21 to 0.88]

10. Secondary Outcome: Change From Baseline in FACT-P:Total Score as a Measure of HRQoL
Description: FACT-P is a 39-item participant questionnaire that measures the concerns of participants with prostate cancer. It consists of 5 sub-scales assessing physical well-being (7 items), social/family well-being (7 items), emotional well-being (6 items), functional well-being (7 items), and prostate-specific concerns (12 items). FACT-P Total Score sums all 5 sub-scales to give a score in the range of 0 to 156, where higher values represent better HRQoL.
Time Frame: as for outcome 9
Population: Analysis was performed on FACT-P population. Number of participants analyzed=participants with evaluable FACT-P Total Score for specified outcome measure. Here, 'n' signifies number of participants with available data for specified category.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Cabazitaxel 20 mg/m^2 | Cabazitaxel 25 mg/m^2
Number analyzed (Participants) | 521 | 495
units on a scale
  Change from baseline at cycle 1 (n =521, 495) | 5.6 [3.43 to 7.78] | 5.75 [3.55 to 7.95]
  Change from baseline at cycle 2 (n = 502, 492) | 5.39 [3.23 to 7.55] | 6.23 [4.05 to 8.42]
  Change from baseline at cycle 3 (n = 459, 452) | 4.39 [2.21 to 6.57] | 6.09 [3.89 to 8.3]
  Change from baseline at cycle 4 (n = 421, 415) | 2.94 [0.73 to 5.14] | 4.2 [1.98 to 6.42]
  Change from baseline at cycle 5 (n = 339, 365) | 1.79 [-0.46 to 4.04] | 3.33 [1.08 to 5.59]
  Change from baseline at cycle 6 (n = 275, 320) | 2.57 [0.26 to 4.88] | 2.35 [0.06 to 4.64]
  Change from baseline at cycle 7 (n = 229, 267) | 2.62 [0.25 to 4.99] | 2.72 [0.38 to 5.06]
  Change from baseline at cycle 8 (n = 196, 226) | 1.35 [-1.08 to 3.78] | 1.98 [-0.42 to 4.37]
  Change from baseline at cycle 9 (n = 164, 172) | 1.1 [-1.4 to 3.6] | 1 [-1.5 to 3.51]
  Change from baseline at cycle 10 (n = 137, 141) | 0.02 [-2.57 to 2.61] | 1.33 [-1.26 to 3.93]
  Change from baseline at Follow-up 1 (n = 137, 153) | -3.1 [-5.69 to -0.51] | -2.09 [-4.65 to 0.46]

11. Secondary Outcome: Percentage of Participants With FACT-P Total Score Response
Description: FACT-P is a 39-item participant questionnaire that measures the concerns of participants with prostate cancer. It consists of 5 sub-scales assessing physical well-being (7 items), social/family well-being (7 items), emotional well-being (6 items), functional well-being (7 items), and prostate-specific concerns (12 items). FACT-P Total Score sums all 5 sub-scales to give a score in the range of 0 to 156, where higher values represent better HRQoL. Responder of FACT-P was defined as at least one occurrence of 7-point improvement from baseline in FACT-P total score during treatment period.
Time Frame: From baseline until DP, start of another anti-cancer therapy, death or study cut-off date (maximum duration: 48 months)
Population: Analysis was performed on FACT-P population. Number of participants analyzed= participants with evaluable FACT-P total score for specified outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cabazitaxel 20 mg/m^2 | Cabazitaxel 25 mg/m^2
Number analyzed (Participants) | 540 | 525
percentage of participants | 57.2 [53.0 to 61.4] | 59.4 [55.2 to 63.6]

12. Secondary Outcome: Time to Definitive Deterioration of Score by 10% From Baseline on FACT-P Sub-Scales
Description: The time to definitive deterioration (10% decrease in score from baseline) was assessed for the individual sub-scales (Physical Well-Being; Social/Family Well-Being; Emotional Well-Being; Functional Well-Being; Prostate-Specific Concerns). Analysis was performed by Kaplan-Meier method.
Time Frame: From baseline until DP, start of another anti-cancer therapy, death or study cut-off date (maximum duration: 48 months)
Population: Analysis was performed on FACT-P population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabazitaxel 20 mg/m^2 | Cabazitaxel 25 mg/m^2
Number analyzed (Participants) | 557 | 543
months
  Physical well-being | 6.6 [5.85 to 7.82] | 8.3 [7.16 to 8.74]
  Social/family well-being | 10.8 [9.26 to 13.37] | 12.4 [8.97 to 13.83]
  Emotional well-being | 9.7 [7.36 to 11.30] | 9.9 [8.54 to 12.52]
  Functional well-being | 6.6 [5.55 to 7.43] | 6.7 [6.01 to 8.34]
  Prostate specific concern | 8.7 [7.62 to 9.66] | 9.7 [8.77 to 10.87]

13. Secondary Outcome: Time to Definitive Deterioration of ECOG PS Score From Baseline
Description: The ECOG PS was used to evaluate participant's DP and the effect of the disease on the participant's activities of daily living. It ranges on the scale from 0-5 (0= normal activity; 1= symptoms but ambulatory; 2= in bed for < 50 % of the time; 3= in bed for > 50% of the time; 4= 100% bedridden; 5= dead). Time to definitive deterioration in ECOG PS score from baseline was defined as a change from 0, 1 to ≥2, or from 2 to ≥3. Analysis was performed by Kaplan-Meier method.
Time Frame: From baseline until death or study cut-off date (maximum duration: 48 months)
Population: Analysis was performed on ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabazitaxel 20 mg/m^2 | Cabazitaxel 25 mg/m^2
Number analyzed (Participants) | 598 | 602
months | 14.9 [11.43 to 23.59] | 14.1 [12.22 to 20.17]

14. Secondary Outcome: Time to Definitive Weight Loss by 5% and 10% From Baseline
Description: Time to definitive weight loss was defined as the time to first occurrence of ≥5% or ≥10% decrease in body weight from baseline. Analysis was performed by Kaplan-Meier method.
Time Frame: From baseline until death or study cut-off date (maximum duration: 48 months)
Population: Analysis was performed on ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabazitaxel 20 mg/m^2 | Cabazitaxel 25 mg/m^2
Number analyzed (Participants) | 598 | 602
months
  Weight Loss by 5% | 10.6 [9.26 to 13.17] | 11.1 [10.12 to 12.42]
  Weight Loss by 10% | NA [12.65 to NA] — The median and upper bound of the confidence interval could not be calculated using the Kaplan-Meier method | 20.3 [14.23 to NA] — The upper bound of the confidence interval could not be calculated using the Kaplan-Meier method

15. Secondary Outcome: Time to First Definitive Consumption of Narcotic Medication
Description: Concomitant medications used were recorded for all participants, and time of first definitive consumption of narcotic medication (if it occurred) was determined. This measure summarizes the time from baseline to first definitive consumption of narcotic medication. Analysis was performed by Kaplan-Meier method.
Time Frame: From baseline until DP, start of another anti-cancer therapy, death or study cut-off date (maximum duration: 48 months)
Population: Analysis was performed on ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabazitaxel 20 mg/m^2 | Cabazitaxel 25 mg/m^2
Number analyzed (Participants) | 598 | 602
months | 2.2 [0.99 to 3.65] | 0.8 [0.30 to 2.20]

16. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Any untoward medical occurrence in a participant who received investigational medicinal product (IMP) was considered an adverse event (AE) without regard to possibility of causal relationship with this treatment. TEAEs: AEs that developed or worsened or became serious during on-treatment period. On-treatment period: The time from the first dose of treatment to 30 days after the last dose of treatment (either Cabazitaxel or Prednisone). A serious adverse event: Any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. Any TEAE included participants with both serious and non-serious AEs. National Cancer Institute Common Terminology Criteria (NCI-CTCAE) version 4.03 (Grade 3 [severe] and Grade 4 [life-threatening]) was used in this study to grade clinical AEs.
Time Frame: From first administration of study treatment until 30 days after the last administration of study treatment (Maximum duration: 48 months)
Population: Safety population included all randomized participants who received at least one dose of the study drug during study treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Cabazitaxel 20 mg/m^2 | Cabazitaxel 25 mg/m^2
Number analyzed (Participants) | 580 | 595
percentage of participants
  Any Grade TEAE | 91.2 | 93.9
  Any Grade 3-4 TEAE | 39.7 | 54.5
  Grade 3-4 TEAE excluding laboratory TEAE | 35.7 | 48.1
  Grade 3-4 TEAE excluding DP TEAEs | 39.0 | 53.9
  Grade 3-4 TEAE excluding laboratory and DP TEAEs | 35.0 | 47.4
  Any Serious TEAE | 30.5 | 43.2
  Any TEAE leading to permanent discontinuation | 16.4 | 19.5

17. Secondary Outcome: Plasma Clearance (CL) for Cabazitaxel
Description: Blood samples for pharmacokinetic (PK) analysis were obtained from a subset of the study participants (approximately 150 participants/group, by protocol) according to a sparse sampling strategy.
Time Frame: Day 1 of Cycle 1: 5 minutes before the end of infusion (EOI), 15 minutes, 1 to 4 hour, 6 to 24 hours, 48 to 168 hour after EOI
Population: Analysis was performed on PK population that included participants who had evaluable PK data. Number of participants analyzed= participants with PK assessment at specified time-points.
Measure: Mean (Standard Deviation); unit: Litre/hour
Arm/Group | Cabazitaxel 20 mg/m^2 | Cabazitaxel 25 mg/m^2
Number analyzed (Participants) | 133 | 166
Litre/hour | 44.832 (15.075) | 49.662 (17.613)

18. Secondary Outcome: Plasma Steady State Volume of Distribution (Vss) for Cabazitaxel
Description: Blood samples for PK analysis were obtained from a subset of the study participants (approximately 150 participants/group, by protocol) according to a sparse sampling strategy.
Time Frame: Day 1 of Cycle 1: 5 minutes before the EOI, 15 minutes, 1 to 4 hour, 6 to 24 hours, 48 to 168 hour after EOI
Population: Analysis was performed on PK population. Number of participants analyzed= participants with PK assessment at specified time-points.
Measure: Mean (Standard Deviation); unit: litre
Groups:
- Cabazitaxel 25 mg/m^2: Cabazitaxel 20 mg/m^2 IV infusion over 1 hour on Day 1 of each 21-day cycle in combination with Prednisone (or Prednisolone) 10 mg orally daily until DP, unacceptable toxicity, participant's refusal of further study treatment or for a maximum of 10 cycles.
Arm/Group | Cabazitaxel 20 mg/m^2 | Cabazitaxel 25 mg/m^2
Number analyzed (Participants) | 133 | 166
litre | 7381.46 (4488.72) | 7040.10 (5133.12)

ADVERSE EVENTS:
Time Frame: All AEs were collected from signature of the informed consent form up to the final visit (48 months) regardless of seriousness or relationship to investigational product.
Description: Reported AEs are TEAEs that is AEs that developed/worsened during the 'on treatment period' (time from first dose of study drug until 30 days after the last administration of study drug). Analysis was performed on safety population.
Arm/Group | Cabazitaxel 20 mg/m^2 | Cabazitaxel 25 mg/m^2
Serious Adverse Events (participants affected / at risk) | 177/580 | 257/595
Other Adverse Events (participants affected / at risk) | 450/580 | 507/595
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cabazitaxel 20 mg/m^2 (N=580) | Cabazitaxel 25 mg/m^2 (N=595)
Abdominal infection (Infections and infestations) | 1 | 0
Amoebic dysentery (Infections and infestations) | 0 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 1 | 1
Cholecystitis infective (Infections and infestations) | 1 | 0
Clostridial infection (Infections and infestations) | 1 | 0
Clostridium bacteraemia (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 2
Febrile infection (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 2 | 0
Listeriosis (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Lymphangitis (Infections and infestations) | 1 | 0
Mastoiditis (Infections and infestations) | 1 | 0
Neutropenic infection (Infections and infestations) | 8 | 17
Neutropenic sepsis (Infections and infestations) | 7 | 14
Pelvic abscess (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 0 | 1
Phlebitis infective (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 6 | 7
Pyelonephritis (Infections and infestations) | 0 | 2
Pyelonephritis acute (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 2
Scrotal infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 5 | 7
Septic shock (Infections and infestations) | 4 | 5
Sinusitis (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 9 | 17
Urinary tract infection bacterial (Infections and infestations) | 1 | 0
Urinary tract infection staphylococcal (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 3 | 2
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 13 | 12
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 10 | 48
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 27
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 3
Drug hypersensitivity (Immune system disorders) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 3 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 1
Ataxia (Nervous system disorders) | 0 | 1
Cerebral haematoma (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Hydrocephalus (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Lumbosacral plexopathy (Nervous system disorders) | 0 | 1
Monoparesis (Nervous system disorders) | 0 | 1
Nerve compression (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Paraparesis (Nervous system disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 6 | 6
Syncope (Nervous system disorders) | 2 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 2 | 3
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardiorenal syndrome (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 3
Embolism venous (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 0 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 | 8
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 5 | 5
Colitis (Gastrointestinal disorders) | 0 | 3
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 13
Diverticular perforation (Gastrointestinal disorders) | 0 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 3
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Enterovesical fistula (Gastrointestinal disorders) | 1 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 1
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 3
Neutropenic colitis (Gastrointestinal disorders) | 0 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 7 | 5
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Gallbladder obstruction (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 8
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 4
Spinal pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 6
Azotaemia (Renal and urinary disorders) | 1 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0
Cystitis noninfective (Renal and urinary disorders) | 1 | 1
Dysuria (Renal and urinary disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 13 | 21
Hydronephrosis (Renal and urinary disorders) | 6 | 7
Renal colic (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 2 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 1 | 0
Urinary bladder toxicity (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 6 | 6
Urinary tract inflammation (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Oedema genital (Reproductive system and breast disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 1
Asthenia (General disorders) | 1 | 4
Catheter site inflammation (General disorders) | 1 | 0
Chest discomfort (General disorders) | 0 | 1
Death (General disorders) | 1 | 1
Device occlusion (General disorders) | 0 | 1
Disease progression (General disorders) | 8 | 13
Fatigue (General disorders) | 1 | 5
General physical health deterioration (General disorders) | 2 | 2
Infusion site extravasation (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 6
Sudden cardiac death (General disorders) | 0 | 1
Sudden death (General disorders) | 1 | 2
Blood creatinine increased (Investigations) | 1 | 2
Neutrophil count decreased (Investigations) | 1 | 1
Transaminases increased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Chemical cystitis (Injury, poisoning and procedural complications) | 0 | 1
Cystitis radiation (Injury, poisoning and procedural complications) | 4 | 4
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 1
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 1
Radiation proctitis (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 0
Urinary anastomotic leak (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cabazitaxel 20 mg/m^2 (N=580) | Cabazitaxel 25 mg/m^2 (N=595)
Urinary tract infection (Infections and infestations) | 33 | 51
Neutropenia (Blood and lymphatic system disorders) | 15 | 40
Decreased appetite (Metabolism and nutrition disorders) | 74 | 108
Dizziness (Nervous system disorders) | 24 | 32
Dysgeusia (Nervous system disorders) | 41 | 63
Peripheral sensory neuropathy (Nervous system disorders) | 38 | 63
Cough (Respiratory, thoracic and mediastinal disorders) | 34 | 35
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 29 | 43
Abdominal pain (Gastrointestinal disorders) | 29 | 48
Constipation (Gastrointestinal disorders) | 102 | 107
Diarrhoea (Gastrointestinal disorders) | 175 | 231
Nausea (Gastrointestinal disorders) | 140 | 188
Stomatitis (Gastrointestinal disorders) | 27 | 30
Vomiting (Gastrointestinal disorders) | 78 | 105
Alopecia (Skin and subcutaneous tissue disorders) | 15 | 36
Arthralgia (Musculoskeletal and connective tissue disorders) | 46 | 37
Back pain (Musculoskeletal and connective tissue disorders) | 63 | 78
Bone pain (Musculoskeletal and connective tissue disorders) | 42 | 42
Pain in extremity (Musculoskeletal and connective tissue disorders) | 30 | 40
Dysuria (Renal and urinary disorders) | 31 | 24
Haematuria (Renal and urinary disorders) | 73 | 108
Asthenia (General disorders) | 88 | 114
Fatigue (General disorders) | 142 | 156
Oedema peripheral (General disorders) | 38 | 53
Pyrexia (General disorders) | 26 | 32
Weight decreased (Investigations) | 24 | 44
Wrong technique in drug usage process (Injury, poisoning and procedural complications) | 2 | 32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.